CLINICAL TRIAL: NCT07276828
Title: Effect Of Autogenic Training On Restless Leg Syndrome And Sleep Disturbance In Hemodialysis
Brief Title: Effect of Autogenic Training on Hemodialysis Patients
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Zainab Gamal Mohamed, Principal Investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P.T.REC/012/006063
Record Dates: First submitted 2025-11-30; First posted 2025-12-11 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-11

CONDITIONS: Hemodialysis Patient; Restless Leg Syndrome (RLS); Fatigue; Sleep Disturbance
MeSH Terms: conditions — Restless Legs Syndrome; Fatigue; Parasomnias | interventions — Autogenic Training

STUDY DESIGN:
Intervention Model Description: Two parallel groups: an intervention group receiving autogenic training and a control group receiving hemodialysis
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental group (autogenic training) (Experimental): 27 patients of both gender will receive the Autogenic Training program in addition to conventional physiotherapy and routin hemodialysis care . The intervention includes guided sessions of autogenic relaxation exercises focusing on breathing regulation, muscle relaxation, and self-induced calming techniques. The sessions will be performed [3] times per week for [8] weeks. The aim of this intervention is to improve sleep quality and reduce symptoms of restless leg syndrome and fatigue in hemodialysis patients.
  Interventions: Behavioral: Autogenic training
- conrol group (Active Comparator): 27 Participants in this group will receive the conventional physiotherapy program routinely provided for hemodialysis patients, with no additional relaxation or autogenic training techniques. This group will be used to compare the effects of adding Autogenic Training to standard physiotherapy.
  Interventions: Other: conventional physical therapy and hemodialysis care

INTERVENTIONS:
Behavioral: Autogenic training — The Autogenic Training Program is a standardized mind-body relaxation technique that uses self-induced verbal formulas and passive concentration to promote autonomic regulation. The intervention includes guided sessions with 6 main exercises , The first exercise aims to relax muscles by repeating a verbal formula, "my right arm is heavy," emphasising heaviness. then feeling warm, initiated by the instruction ''my right arm is warm'', followed by cardiac activity using the formula ''my heartbeat is calm and regular''. Then follows passive concentration on the respiratory mechanism with the formula ''it breathes me'', then on warmth around the abdominal region with ''my solar plexus is warm'' and finally on coolness in the cranial region with ''my forehead is cool and clear'' . Participants will receive supervised training sessions followed by home practice instructions to enhance relaxation response and reduce physiological stress. in addition to conventional physiotherapy program
  Arms: experimental group (autogenic training)
Other: conventional physical therapy and hemodialysis care — control group will receive a conventional physiotherapy program that includes stretching exercises, strengthening exercises, range-of-motion training, and standard therapeutic procedures routinely used for patients with similar conditions. The sessions will follow a structured protocol delivered by a physiotherapist, without including any relaxation or autogenic training components.
  Arms: conrol group

SUMMARY:
goal of this interventional study to investigate the effect of autogenic training on sleep disturbance , restless leg syndrome and fatigue on hemodialysis patient Is there any significant effect of autogenic training on restless leg syndrome, sleep disturbance and fatigue in patients with hemodialysis?

The intervention will include structured autogenic training sessions, and outcomes such as sleep quality and RLS severity and fatigue will be evaluated after 8 weeks of autogenic training on hemodialysis patients .

DETAILED DESCRIPTION:
Hemodialysis patients always face various problems such as fatigue and sleep disturbance due to the chronic nature and side effects of hemodialysis, which negatively affect their quality of life A variety of treatment regimens can be chosen to initially relieve symptoms of patients currently with RLS and fatigue, among available regimes, pharmacological treatments are mainly selected for cases with severe RLS, which, at times, lead to serious complications It is hypothesized that these patients, according to the above implications, require a treatment suitable to their somatopsychic necessity, that autogenic training should perform being a method of choice for these types of issues Few clinical trials have examined the efficacy of autogenic training in patients undergoing hemodialysis that suffering from fatigue, restless syndrome and sleep disturbance, this approach could be incorporated into routine care protocols, enhancing patient comfort, promoting self-management, and reducing reliance on medications and their complications.

ELIGIBILITY:
Inclusion Criteria

* Age between 45 and 55 years.
* Body Mass Index (BMI) between 25.0 and 29.9 kg/m².
* Clinically and medically stable.
* On hemodialysis for at least 6 months prior to enrollment.
* Diagnosed with chronic kidney disease (CKD), defined by one or more of the following:

Evidence of kidney damage (e.g., albuminuria), or

Decreased kidney function with glomerular filtration rate (GFR) < 60 mL/min/1.73 m² for ≥ 3 months, irrespective of clinical diagnosis.

*Systolic blood pressure < 140 mmHg, diastolic blood pressure < 90 mmHg, and heart rate < 80 bpm.

Exclusion Criteria

Uncontrolled pulmonary disease.

Severe vascular complications (e.g., critical limb ischemia).

Unstable angina.

Uncontrolled cardiac arrhythmia.

Decompensated heart failure.

Cognitive impairment.

Participants who miss more than two weeks of the program or request termination.

Ages: 45 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 54 (Estimated)
Dates: Start 2025-12-15 (Estimated); Primary Completion 2027-03-15 (Estimated); Study Completion 2027-05-15 (Estimated)

PRIMARY OUTCOMES:
Dialysis adequacy | 8 weeks
  Dialysis adequacy will be assessed using URR (Urea Reduction Ratio) measured pre- and post-intervention to determine the effectiveness of the treatment in improving hemodialysis efficiency."

SECONDARY OUTCOMES:
sleep disturbance | 8 weeks
  Sleep disturbance will be assessed using the Pittsburgh Sleep Quality Index (PSQI) questionnaire. Changes in total score and specific subcomponents (sleep latency, sleep duration, sleep efficiency, sleep disturbances, use of sleep medication, and daytime dysfunction) will be measured before and after the intervention.", each rated on a 0 to 3 scale, with higher scores implying greater difficulties. PSQI < 5 indicates good sleep quality; PSQI ≥ 5
restless leg syndrome | 8 weeks
  Restless Leg Syndrome will be assessed using the International Restless Legs Syndrome Study Group (IRLSSG) rating scale. Severity and frequency of symptoms will be measured at baseline and after the intervention to evaluate improvement IRRLSSG severity questionnaire consisting of ten questions . In this questionnaire, all the answers have a score ranging from 0 (corresponding to "none") to 4 (corresponding to "very large") and the final score represents the sum of the answers of the ten questions, 0 to 10 points, light; 11 to 20 points, moderate; 21 to 30 points, serious; and 31 to 40 points, very serious
fatigue | 8 weeks
  Fatigue will be assessed using the Fatigue assessment Scale (FAS). Changes in severity and impact on daily activities will be measured at baseline and after the intervention.
  It is a standardized 10-item Likert scale ranging from 1 ("never") to 5 ("always"). It is used to assess the symptoms of fatigue. The tool reliability was 0.96. Each item of the FAS is answered using a five-point scale. Total scores range from 10 to 50, where score 10 indicates the mildest level of fatigue and score 50 denotes the highest level of fatigue among the participants

CONTACTS AND LOCATIONS:
Locations (1):
- Faculity of physical therapy, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No